CLINICAL TRIAL: NCT03758430
Title: Technology-supported, Meal-centric, Insulin Dosing for Optimized Post-prandial Glucose Control
Brief Title: A Study of Technology to Improve Glucose Control in Participants With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Joslin Diabetes Center (Other)
Responsible Party: Sponsor
Other Study IDs: 17111; F3Z-MC-IORA (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Fitness Trackers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Combined Diabetes Management Data: Participants with type 1 diabetes will use a meal tagging application (app) and fitness tracker. They will upload these data to a web portal where they will be matched with data from their continuous glucose monitor and insulin pump. Combined data will be used for diabetes management.
  Interventions: Other: Meal-Tagging App; Device: Fitness Tracker

INTERVENTIONS:
Other: Meal-Tagging App — Meal tagging app to capture frequently eaten meals and test meals for 16 weeks.
Device: Fitness Tracker — Fitness tracker will be worn around the clock for 16 weeks.

SUMMARY:
The main purpose of this study is to determine whether combining meal, glucose, and insulin data in a web-based system will improve management of type 1 diabetes (T1D). No study drug will be given. The study will last about 18 weeks.

ELIGIBILITY:
Inclusion Criteria:

* T1D by clinical diagnosis for > 3 years
* Insulin pump use > 3 months: must use one of the following pump types: Animas Ping and Vibe, Insulet Omnipod, Medtronic 523/723 and 530G, Tandem t:slim and t:flex
* Continuous Glucose Monitor (CGM) > 3 months and current use of Dexcom G5 at least 6 out of 7 days per week
* HbA1c 7.0-9.5%
* Must have iPhone (meal-tagging app has been built on iOS)
* Personal computer for uploading of pump and CGM devices
* Willingness to follow study protocol including tagging food data
* Comfort speaking, reading, and writing English

Exclusion Criteria:

* Individuals currently using a hybrid closed-loop system (e.g., Medtronic 670G)
* Individuals planning to follow a specific diet plan for weight loss
* Inability to consume "common meals"
* Gastroparesis;
* Eating disorder
* Evidence of missed insulin meal-time insulin boluses on pump download
* Use of medications that can affect blood glucose levels (such as SGLT inhibitors, steroid, beta agonists)
* Use of medications that affect gastric emptying (such as GLP agonists, pramlinitide)
* Alcohol abuse
* Pre-conception, pregnancy, or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with T1D
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2020-08-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Week 16 in Hemoglobin A1c (HbA1c) | Baseline to Week 16
  Change from Baseline to Week 16 in HbA1c

SECONDARY OUTCOMES:
Change from Baseline to Week 16 in Post-Prandial Glucose Concentrations Following Commonly Eaten Meals | Baseline to Week 16
  Change from Baseline to Week 16 in Post-Prandial Glucose Concentrations Following Commonly Eaten Meals

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No